CLINICAL TRIAL: NCT03426579
Title: Correlation Between Sedation Depth Monitoring and Reflexes During Intravenous Anesthesia With Dexmedetomidine and Remifentanil in Children Undergoing Direct Laryngoscopy for Surgical Procedures
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Joke De Wachter, data manager, University Hospital, Antwerp
Other Study IDs: 17/31/360
Record Dates: First submitted 2017-10-23; First posted 2018-02-08 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Laryngoscopy; Child; Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Reliability of NeuroSENSE ®in children: Children scheduled for direct laryngoscopy with surgical intervention the reliability of NeuroSENSE ®monitoring will be evaluated
  Interventions: Device: NeuroSENSE ®in children

INTERVENTIONS:
Device: NeuroSENSE ®in children — Before induction of anesthesia NeuroSENSE ® monitoring will be applied to all subjects.General anesthesia with dexmedetomidine and remifentanil is titrated based on the evaluation of respiratory clinical signs (cough, spasm, movement) and immobility of the vocal cords. The anesthesiologist performing anesthesia will be blinded for the Wavelet-based Anesthetic Value for Central Venous System (WAVCNS) index assessed by NeuroSENSE ® and will adjust dexmedetomidine according to clinical signs, which is standard of care. Retrospectively data obtained by NeuroSENSE ® will be compared to evaluate whether they are useful in predicting upcoming unwanted airway reflexes.

SUMMARY:
This study evaluates the correlation between sedation depth monitoring obtained by NeuroSENSE ® NS 701 Monitor and reflexes during intravenous anesthesia in children undergoing direct laryngoscopy for surgical procedures.

DETAILED DESCRIPTION:
Direct laryngoscopy for invasive procedures in children is performed under general anesthesia with spontaneous or controlled ventilation.Preventing under-or over-sedation and titration of sedation according to patient needs with spontaneous ventilation is a real challenge. It is common practice that dexmedetomidine and remifentanil are titrated based on the evaluation of respiratory clinical signs (cough, spasm, movement) and immobility of the vocal cords.NeuroSENSE ®NS 701 Monitor( NeuroWave Systems incorporated - Cleveland Heights,OH) is a sedation depth monitor that uses automated electroencephalogram quantification. It provides information about depth of anesthesia before change of clinical signs.The primary reason for WAVCNS monitoring is to prevent under-or over-sedation, to titrate sedation according to patient needs. NeuroSENSE ® is validated for monitoring sedation depth in adults but not in children. The Wavelet-based Anesthetic Value for Central Venous System (WAVCNS) index calculated by this monitor is scaled into the 100-0 range, where 100 denotes a brain state consistent with an awake patient and a 0 denotes a total and prolonged absence of cortical activity. The recommended WAVCNS index range for general anesthesia is between 40-60 as within this range there is very low probability of a patient being either awake or in deep anesthetic state. The validated use of a sedation depth monitor in children, who are at risk for medication overdosage or airway spasm by underdosing sedatives, could be a major advantage. In this trial ten children scheduled for direct laryngoscopy with surgical intervention will be enrolled after obtaining written informed consent of their parents or legal guardian.The NeuroSENSE ®monitor will be installed previous to anesthesia induction. The attending anesthesiologist is instructed to guide titration of dexmedetomidine/ remifentanil according to clinical signs, which is standard of care. He is blinded for the NeuroSENSE ® monitor.Induction of anesthesia will be done with sevoflurane an a bolus of dexmedetomidine 4 microgram/kilogram will be administered. Maintenance of anesthesia will be accomplished with dexmedetomidine infused at 2 microgram/kilogram/hour and adjusted to clinical needs with top up bolus dexmedetomidine of 0.5 microgram/kg/hour. Remifentanil will be infused at 0.3 mcg/kg/min and adjusted to clinical needs to 0.5 mcg/kg/min. Before start of surgery, on visualising the vocal cords 1 spray of 10 percent lidocaine is delivered to anesthetize the vocal cords. all children receive pharyngeal tube for oxygen supplementation. Spontaneous ventilation will be maintained. In case of laryngospasm and desaturation, propofol will be used as rescue medication. After surgery all children will be monitored on Intensive Care or Post Anesthetic Care Unit as standard of care. Heart rate, non-invasive blood pressure, pulse oxygen saturation, respiratory rate will be recorded at Innovian (Drager Medical Systems, Andover, USA) Induction time, adverse events, incidence of leg movements during anesthesia, cough, postoperative awakening and recovery time will be assessed.Surgery satisfaction will be assessed using score 1 is extremely dissatisfied; 2 is not satisfied but able to manage; 3 is extremely satisfied. At end of surgery total cumulative dose of dexmedetomidine and remifentanil will be calculated. Results from NeuroSENSE ® are extracted as raw data from the device.

ELIGIBILITY:
Inclusion Criteria:

scheduled for elective direct laryngoscopy with surgical intervention, written informed consent of their parents or legal guardian.

Exclusion Criteria:

refusal of informed consent, known allergy for dexmedetomidine or remifentanil at start of anesthesia pulse oxygen saturation (SaO2) lower than 85%

Ages: 1 Month to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children scheduled for direct laryngoscopy with surgical intervention
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2017-10-23 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
predictability of NeuroSENSE ® in upcoming unwanted airway reflexes | during surgery
  Define whether the NeuroSENSE ® provides information before upcoming clinical signs about under- or over-sedation defined as cough, laryngospasm, apnea or desaturation

SECONDARY OUTCOMES:
Incidence of leg movement | During surgery
  Incidence of any lower limb movement during anesthesia
Total cumulative dose of dexmedetomidine | From induction of anesthesia till extubation with a maximum up to 4 hours after intubation
  Total dose of dexmedetomidine during anesthesia in microgram
Total cumulative dose of remifentanil | From induction of anesthesia till extubation with a maximum up to 4 hours after intubation
  Total dose of remifentanil during anesthesia in microgram
Postoperative awaking time | Time between end of surgery and opening of the eyes in minutes, up to a maximum of 30 minutes
  Time between end of surgery and addressability of the patient in minutes

CONTACTS AND LOCATIONS:
Overall Officials: Vera Saldien, Principal Investigator — University Hospital, Antwerp
Locations (1):
- University hospital Antwerp, Edegem, Antwerp, Belgium